CLINICAL TRIAL: NCT02129179
Title: The Effect of Glucagon-Like Peptide-1 (GLP-1) on Pulmonary Vascular Resistance (PVR) in Patients With Heart Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PO1860
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Glucagon-Like Peptide 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GLP-1 (Experimental)
  Interventions: Drug: Glucagon-Like Peptide 1

INTERVENTIONS:
Drug: Glucagon-Like Peptide 1

SUMMARY:
This study aims to assess the effect of glucagon-like peptide-1 on cardiac output and transpulmonary gradient in patients undergoing right heart catheterisation for clinical reasons.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Able to give informed consent
* On the waiting list for heart transplant
* Left Ventricular Dysfunction awaiting catheterisation

Exclusion Criteria:

* Nicorandil, glibenclamide, Dipeptidyl Peptidase-4 inhibitor, Glucagon-Like Peptide-1 receptor agonist or insulin
* Women of child bearing age and breast feeding women
* Cardiac pacemaker or other implanted metallic device
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Pulmonary Vascular Resistance with Glucagon-Like Peptide-1 | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Papworth Hospital NHS Foundation Trust, Papworth Everard, United Kingdom

REFERENCES:
- [Derived] Clarke SJ, Pettit S, Giblett JP, Zhao T, Kydd AC, Albrechtsen NJW, Deacon CF, Parameshwar J, Hoole SP. Effects of Acute GLP-1 Infusion on Pulmonary and Systemic Hemodynamics in Patients With Heart Failure: A Pilot Study. Clin Ther. 2019 Jan;41(1):118-127.e0. doi: 10.1016/j.clinthera.2018.11.013. Epub 2018 Dec 28. PMID 30598343